CLINICAL TRIAL: NCT05254626
Title: Efficacy and Safety of Dapagliflozin Compared to Pioglitazone in Diabetic and Non-diabetic Patients with Non-alcoholic Steatohepatitis
Brief Title: Efficacy and Safety of Dapagliflozin in Patients with Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nirmeen Ahmed Sabry, Professor Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (3148)
Record Dates: First submitted 2021-12-01; First posted 2022-02-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Dapagliflozin; SGLT2 inhibitors; NASH; Efficacy; Safety; Liver biopsy; Pioglitazone; Fatty Liver; NAFLD activity score
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — dapagliflozin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diabetic Group 1 (Experimental): 25 diabetic patients will be prescribed on dapagliflozin 10 mg - once daily (OD) - to be taken orally (PO) for 24 weeks
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Diabetic Group 2 (Active Comparator): 25 diabetic patients will be prescribed on Pioglitazone 30 mg - once daily (OD) - to be taken orally (PO) for 24 weeks
  Interventions: Drug: Pioglitazone 30 mg
- Non-diabetic Group 1 (Experimental): 25 non-diabetic patients will be prescribed on dapagliflozin 10 mg - once daily (OD) - to be taken orally (PO) for 24 weeks.
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Non-diabetic Group 2 (Active Comparator): 25 non-diabetic patients will be prescribed on Pioglitazone 30 mg - once daily (OD) - to be taken orally (PO) for 24 weeks
  Interventions: Drug: Pioglitazone 30 mg

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Dapagliflozin 10 mg, administered orally and to be prescribed for diabetic and non-diabetic patients with NASH for 24 weeks; in comparison to pioglitazone.
  Arms: Diabetic Group 1; Non-diabetic Group 1
Drug: Pioglitazone 30 mg — Pioglitazone 30 mg, administered orally and to be prescribed for diabetic and non-diabetic patients with NASH for 24 weeks; as an active control and standard of care treatment.
  Arms: Diabetic Group 2; Non-diabetic Group 2

SUMMARY:
Patients with non-alcoholic fatty liver disease (NAFLD) are at increased risk of more aggressive liver disease; non-alcoholic steatohepatitis (NASH) and at a higher risk of death from cirrhosis, hepatocellular carcinoma and cardiovascular diseases. NAFLD is spreading as an epidemic in patients with metabolic syndrome. Its components include obesity, type 2 diabetes mellitus (T2DM) and dyslipidemia. The prevalence of NAFLD is likely to increase resulting in tremendous clinical, social and economic burdens. Unfortunately, there is no approved medication to treat patients with NASH-induced advanced fibrosis. Weight management is the first line of NASH treatment even in non-obese patients with at least 7% reduction of patient's weight. However, NASH patients need pharmacological treatment. Sodium glucose co-transporter (SGLT2) inhibitors demonstrated favorable effects on NAFLD without weight gain as an adverse event proposed by pioglitazone used for the same indication. SGLT2 inhibitors are able to reduce fatty liver content, as assessed by different imaging techniques, and improve biological markers of NAFLD, especially serum liver enzymes, in patients with or without T2DM. In addition, there are emerging data to suggest a mechanism beyond the reduction of body weight and hyperglycemia in patients with or without diabetes.

This study aims to evaluate the efficacy and safety of SGLT2 inhibitors in NASH patients in comparison to pioglitazone.

This is a randomized prospective parallel study, where all patients presented with NASH to the outpatient clinic in the National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt; will be screened for specific inclusion and exclusion criteria. Diabetic and non-diabetic patients will be randomly assigned to receive one of two treatment modalities. The first arm will be the NASH patients receiving dapagliflozin and the second arm will be the NASH patients receiving pioglitazone for 24 weeks. Each group will have an equal number of diabetic and non-diabetic patients.

All patients will be assessed for body composition, serum creatinine level, fasting blood glucose level, HbA1C, markers of insulin resistance (HOMA-IR), complete blood count, serum liver function tests, and NAFLD fibrosis score (NAS). Liver biopsy will be performed at baseline and at the end of the study and the total NAS score will be calculated. All patients will be assessed for any adverse drug reactions, and for their adherence by pill count method. Also, quality of life will be assessed for all patients using previously designed and validated questionnaire called Chronic Liver Disease Questionnaire (CLDQ).

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65 years.
* Liver biopsy confirming NASH within 6 months.
* For diabetic patients, the patients should be with stable glycemic control defined as HbA1C <10%.

Exclusion Criteria:

* Active viral hepatitis (HBV, HCV).
* Child Pugh B or C cirrhosis.
* Alcohol consumption in the past six months.
* A history of alcoholic liver disease.
* Secondary causes of steatohepatitis.
* Autoimmune hepatitis.
* Celiac disease.
* Hemochromatosis or Wilson's disease.
* Drug induced liver injury (DILI) or patient with history of taking medication(s) that may cause fatty liver (e.g., tamoxifen, valproic acid, amiodarone, methotrexate, steroids, oral contraceptives).
* Obstructive biliary disease.
* Serum alanine aminotransferase (ALT) more than 2.5 folds of UNL.
* History of serious hypersensitivity to dapagliflozin or pioglitazone or any component of the formulation.
* Pregnancy and breastfeeding.
* Renal impairment (eGFR <45 mL/minute/1.73 m2), end-stage renal disease (ESRD), or patients on dialysis.
* Having any medical condition that would affect metabolism (i.e., known hyperthyroidism or hypothyroidism).
* Hypopituitarism.
* Patients with Type 1 diabetes.
* Starvation.
* Serious medical disease with likely life expectancy less than 5 years.
* Participation in other clinical trial in the 30 days before enrollment.
* Patients who are unwilling or unable to give informed consent.
* Patients on statins.
* Heart failure defined as New York Heart Association (NYHA) class III or IV.
* Recent initiation or change of antidiabetic drugs that influence liver fat including thiazolidinediones, glucagon like peptide 1 receptor agonists or any SGLT2 inhibitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Histological Features (Liver Biopsy) | Baseline and 24th week
  Change from baseline of NAFLD Activity Score (NAS) and other histological features. NAS score will be assessed using the NASH Clinical Research Network (NASH CRN) scoring system. NAS score ranges from 0 to 8 and the higher score towards 8 means worse outcome.

SECONDARY OUTCOMES:
NAFLD fibrosis score | Baseline and 24th week
  Change in NAFLD fibrosis score (NFS). The score ranges from < -1.45 (no significant fibrosis) to > 0.67 (significant fibrosis). The higher score means worse outcome.
Fibrosis Index Based on 4 factors | Baseline and 24th week
  Change in Fibrosis Index Based on 4 factors (FIB-4). The score ranges from < 1.45 (minimal to no fibrosis) to > 3.4 (advanced fibrosis). The higher score means worse outcome.
Fibro-controlled attenuated parameter (fibro CAP) | Baseline and 24th week
  Improvement of fibro-controlled attenuated parameter (fibro CAP)
Serum Alanine Transaminase level (ALT) | Baseline, 12th and 24th week
  Change in ALT serum level as inflammatory markers of NASH
Serum Aspartate Aminotransferase level (AST) | Baseline, 12th and 24th week
  Change in AST serum level as inflammatory markers of NASH
Serum Alkaline Phosphatase level (ALP) | Baseline, 12th and 24th week
  Change in ALP serum level as inflammatory markers of NASH
Serum Gamma-glutamyl Transferase level (GGT) | Baseline, 12th and 24th week
  Change in GGT serum level as inflammatory markers of NASH
Serum total and direct bilirubin. | Baseline, 12th and 24th week
  Change in levels of serum total and direct bilirubin.
Waist circumference | Baseline, 3rd, 6th, 12th, 18th and 24th week
  Change in waist circumference
Body weight | Baseline, 3rd, 6th, 12th, 18th and 24th week
  Change in body weight
Lipid profile | Baseline, 12th and 24th week
  Change in serum lipids
Glycated hemoglobin (HbA1C) | Baseline, 12th and 24th week
  Change in HbA1C level for patients with T2DM
Fasting blood glucose level | Baseline, 3rd, 6th, 12th, 18th and 24th week
  Change in fasting blood glucose for patients with T2DM
Insulin resistance (HOMA-IR) | Baseline, 12th and 24th week
Quality of life Questionnaire (quality of life assessment) | Baseline and 24th week
  Change in health-related quality of life scores using chronic liver disease questionnaire (CLDQ)
Drugs adverse events | Baseline, 3rd, 6th, 12th, 18th and 24th week
  Assessment of safety by reporting any adverse events

OTHER OUTCOMES:
Serum creatinine | Baseline, 3rd, 6th, 12th, 18th and 24th week
Estimated glomerular filtration rate (eGFR) | Baseline, 3rd, 6th, 12th, 18th and 24th week

CONTACTS AND LOCATIONS:
Overall Officials: Nirmeen A. Sabry, Principal Investigator — Clinical Pharmacy Department - Faculty of Pharmacy - Cairo university
Locations (1):
- National Hepatology and Tropical Medicine Research Institute, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel Monem MS, Adel A, Abbassi MM, Abdelaziz DH, Hassany M, Raziky ME, Sabry NA. Efficacy and safety of dapagliflozin compared to pioglitazone in diabetic and non-diabetic patients with non-alcoholic steatohepatitis: A randomized clinical trial. Clin Res Hepatol Gastroenterol. 2025 Mar;49(3):102543. doi: 10.1016/j.clinre.2025.102543. Epub 2025 Jan 29. PMID 39884573